CLINICAL TRIAL: NCT06815172
Title: PARA (Pancreatic Adenocarcinoma Etiology: Role of Asbestos): Study of Risk Factors for Exocrine Pancreatic Neoplasms.
Brief Title: PARA (Pancreatic Adenocarcinoma Etiology: Role of Asbestos) Study of Risk Factors for Exocrine Pancreatic Neoplasms.
Acronym: PARA
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: PARA; RC-2022-2773381 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2025-01-10; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: asbesto; cancer; risk factor; pancreatic adenocarcinoma
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — tissue sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: 100 subjects will be patients seen on an outpatient basis and suffering from pancreatic adenocarcinoma with histological confirmation, contacted both during hospitalization and during outpatient access or in day service
- Group B: 400 subjects will be patients already included as controls in the CARA study (Cholangiocarcinoma Aetiology: Role of Asbestos - code 111/2013/UOSS evaluated in the meeting of the Ethics Committee of 19/11/2013) admitted to the Polyclinic in the ophthalmology, urology and gynecology departments not affected by the pathology under study, nor by pathologies associated with exposure to asbestos.

SUMMARY:
The primary objective of the study will be to evaluate the possible association between asbestos exposure (occupational, paraoccupational, environmental and non-occupational) and pancreatic adenocarcinoma. The data collected will be used to generate specific hypotheses on the possible environmental and occupational determinants of the disease.

The study aims to evaluate:

1. To evaluate the exposure to asbestos occurred during life, through the use of a standardized questionnaire to be administered to incident cases (newly diagnosed) of histologically diagnosed pancreatic adenocarcinoma afferent to the Medical Oncology Unit Prof. Ardizzoni in Group A, the exposure to asbestos occurred during the course of life;
2. To produce quantitative estimates of the risk of pancreatic adenocarcinoma associated with asbestos exposure.

2.3. To evaluate the presence of asbestos fibers directly on histological sections of pancreatic cancer of patients exposed to asbestos and undergoing surgery.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) ranks fourth among the causes of cancer death in Western countries, with an incidence almost comparable to mortality. The only therapeutic option with curative intent is surgery, but about 80% of subjects diagnosed with this neoplasm are not candidates for surgery due to the presence of distant metastases (stage IV according to the TNM system) or in the case of locally advanced disease (stage III), with an overall survival at 5 years of less than 10%.

Numerous risk factors have been related to the genesis of PDAC both environmental and genetic.

Environmental factors include cigarette smoking, dietary habits such as high intake of animal proteins and fats, high salt consumption, dehydrated foods, smoked meat, fried foods and smoked sugar, obesity, consumption of high amounts of alcohol, occupational exposure to chlorinated hydrocarbons, chronic pancreatitis and type II diabetes mellitus.

However, most of them are non-specific and there is often no concordance between the different studies conducted to evaluate them.

The role of asbestos exposure as an environmental risk factor in the etiopathogenesis of pancreatic cancer has been poorly investigated to date and with discordant results.

However, as previously demonstrated, asbestos, once inhaled, can enter the lymphatic circulation and therefore the bloodstream by accumulating in the tissues. In particular, a deposit of asbestos fibers in the liver has been demonstrated with the possibility of triggering chronic inflammatory mechanisms underlying the carcinogenic process. Similarly to what has already been demonstrated on the association between occupational exposure to asbestos and the risk of intrahepatic cholangiocarcinoma, this observational study aims to evaluate a possible correlation between this environmental risk factor and pancreatic cancer.

Materials and methods A prospective non-pharmacological single-center observational study will be carried out.

A total of 500 subjects will be involved between Group A and Group B, distributed as follows:

* 100 subjects of Group A will be patients seen on an outpatient basis and suffering from pancreatic adenocarcinoma with histological confirmation, contacted both during hospitalization and during outpatient or day service access;
* 400 subjects of Group B will be patients already included as controls in the CARA study (Cholangiocarcinoma Aetiology: Role of Asbestos - code 111/2013/UOSS evaluated in the meeting of the Ethics Committee of 19/11/2013) admitted to the Polyclinic in the ophthalmology, urology and gynecology departments not affected by the pathology under study, nor by pathologies associated with exposure to asbestos.

Upon obtaining informed consent, all subjects in Group A will be administered a standardized questionnaire (once per patient), containing questions from the ReNaM questionnaire (National Mesothelioma Registry), the work history of the subjects and some questions related to known risk factors.

Descriptive population statistics will be presented, stratifying according to case or control status. To estimate the strength of the association between asbestos exposure and pancreatic cancer risk, uni- and multivariate logistic models will be conducted.

On 30 cases subjected to the ReNaM questionnaire, the presence of asbestos fibers directly on histological sections of pancreatic cancer, obtained following surgical resection for curative therapeutic purposes according to the standard of care, will be evaluated.

Samples will be evaluated using light microscopy and scanning electron microscopy with attached chemical microprobe to highlight the presence of fibers within the tumor tissue.

ELIGIBILITY:
Group A

Inclusion Criteria:

1. Incident cases (new diagnosis) of histologically diagnosed pancreatic adenocarcinoma afferent to the Medical Oncology Unit Prof. Ardizzoni
2. Age 30-90 years
3. Ability to complete the questionnaire
4. Ability to read and understand Italian
5. Signing the informed consent form

Exclusion Criteria:

1. Prevalent cases of the pathology under study

Group B

Inclusion Criteria:

1. Patients admitted to the S.Orsola-Malpighi Polyclinic in the ophthalmology, gynecology and urology departments with a diagnosis of cataracts, uterine fibroids and prostate adenoma previously included in the CARA study.
2. Age 30-90 years
3. Ability to complete the questionnaire
4. Ability to read and understand Italian
5. Signing the informed consent form

Exclusion Criteria:

1. Patients with pancreatic adenocarcinoma
2. Patients with a history of malignant neoplastic pathologies
3. Patients suffering from diseases associated with exposure to asbestos: pleuropatias (parietal plaques, diffuse visceral thickening, recurrent effusions and round atelectasis) and pulmonary diseases (alveolitis and asbestosis)
4. Patients in danger of life or hospitalized waiting to undergo surgery for pathologies other than those of inclusion

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The maximum duration of the enrollment period will be 32 years, in which 100 participants from Group A and 400 participants from Group B (previously enrolled in the CARA study (Cholangiocarcinoma Aetiology: Role of Asbestos - Study of risk factors of biliary neoplasms) with code 111/2013/UOSS evaluated in the meeting of the Ethics Committee on 19/11/2013 will be recruited.
  In each case, four hospital checks will be matched, in frequency matching by sex and five-year age group. The choice of this ratio between Group A and Group B (1:4) is justified by the desire to maximize the statistical power of the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
primary objective | From enrollment to the administration of the standardized questionnaire (once per patient), containing questions from the ReNaM (National Mesothelioma Registry) for up to 60 days.
  The primary objective of the study will be to evaluate the possible association between asbestos exposure (occupational, paraoccupational, environmental and non-occupational) and pancreatic adenocarcinoma. The data collected will be used to generate specific hypotheses on the possible environmental and occupational determinants of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: GIOVANNI BRANDI, MD, PHD, Principal Investigator — University of Bologna
Locations (1):
- Irccs Aoubo, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided